CLINICAL TRIAL: NCT07059884
Title: Distance-Based Exercise to Preserve Function and Prevent Disability
Acronym: DEFEND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: A222302
Record Dates: First submitted 2025-06-23; First posted 2025-07-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Localized Malignant Solid Neoplasm
MeSH Terms: interventions — Telemedicine; Accelerometry; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (DEFEND) (Experimental): Patients complete supervised TH exercise sessions consisting of progressive resistance exercise BIW and complete unsupervised aerobic exercise sessions over 30 minutes TIW until the end of SOC chemotherapy or up to a total of 6 months, whichever comes first, in the absence of disease progression or unacceptable toxicity. Patients also receive adjustable-weight dumbbells on study and wear an accelerometer throughout the study.
  Interventions: Other: Exercise intervention; Other: Telemedicine; Other: Aerobic Exercise Intervention; Other: Dumbbell Exercise Intervention; Procedure: Accelerometry; Other: Questionnaire Administration; Other: Interview; Other: Electronic Health Record Review

INTERVENTIONS:
Other: Exercise intervention — Complete supervised TH progressive resistance exercise sessions
Other: Telemedicine — Complete supervised TH progressive resistance exercise sessions
  Other Names: Telehealth
Other: Aerobic Exercise Intervention — Complete unsupervised aerobic exercise sessions
Other: Dumbbell Exercise Intervention — Receive adjustable-weight dumbbells
Procedure: Accelerometry — Wear accelerometer
Other: Questionnaire Administration — Ancillary studies
Other: Interview — Ancillary studies
Other: Electronic Health Record Review — Ancillary studies

SUMMARY:
This clinical trial studies whether an exercise program can be successfully delivered to patients receiving treatment for cancer through virtual sessions and allow patients to exercise in their own home. Treatments for cancer can cause side effects such as fatigue and loss of strength. These side effects can make it difficult to work, take care of family, and do other things the patient wants to do. Preliminary research shows that exercise can help prevent some of these side effects, but it can be more difficult to start an exercise program when a patient is receiving cancer treatment. The exercise program in this study is delivered through telehealth (TH) video calls. The TH sessions are delivered by trained staff that supervise resistance exercises. The trained staff also provide guidance to the patient on completing unsupervised aerobic sessions on their own. This may be a successful way to deliver an exercise program and make it easier for cancer patients to exercise in their own home during treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the feasibility of implementing a virtual exercise intervention trial in a diverse cohort of cancer patients undergoing chemotherapy.

SECONDARY OBJECTIVE:

I. To establish feasibility of enrolling and retaining a diverse patient population.

EXPLORATORY OBJECTIVES:

I. Evaluate changes in 6 Minute Walk Test (6MWT) distance in the study population between baseline and the post-chemotherapy time point.

II. Evaluate changes in grip strength in the study population between baseline and the post-intervention time point.

III. Evaluate objective (accelerometer) and self-reported changes (7-Day Physical Activity Recall Interview) in physical activity in the study population between baseline and the post-intervention time point.

IV. Explore the relationship between the predicted 6MWT and the baseline 6MWT. V. Explore changes in patient reported outcomes between baseline, end of intervention, and 3-months post intervention in the study population.

VI. Explore employment status over time in the study population.

OUTLINE:

Patients complete supervised TH exercise sessions consisting of progressive resistance exercise twice a week (BIW) and complete unsupervised aerobic exercise sessions over 30 minutes three times per week (TIW) until the end of standard of care (SOC) chemotherapy or up to a total of 6 months, whichever comes first, in the absence of disease progression or unacceptable toxicity. Patients also receive adjustable-weight dumbbells on study and wear an accelerometer throughout the study.

After completion of study intervention, patients are followed up at 4 weeks and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Participants must have histologically confirmed cancer
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Participants must be initiating outpatient cytotoxic chemotherapy for curative intent (for any malignancy) of at least 10 weeks duration (with or without concurrent radiation, immunotherapy, or other targeted therapy). Patients must be enrolled and baseline measures collected on or before administration of their second cycle of cytotoxic therapy. Patients receiving outpatient cytotoxic chemotherapy for curative intent in the neoadjuvant or adjuvant setting for solid tumors are eligible. Patients receiving outpatient cytotoxic chemotherapy given for curative intent for hematologic malignancies, as well as patients receiving definitive chemoradiation for solid tumors, are also eligible. Regimens of immunotherapy or monoclonal antibodies ONLY are not eligible
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Age 18-64 years
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Patients cannot have metastatic cancer
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Patients cannot have documentation in the medical record of severe cardiovascular, respiratory or musculoskeletal disease or joint problems that preclude moderate physical activity. Examples would include unstable angina, recent myocardial infarction, oxygen-dependent pulmonary disease, and osteoarthritis requiring imminent joint replacement. Moderate arthritis that does not preclude physical activity is not a reason for ineligibility
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Patients cannot be pregnant, because this study involves remotely delivered exercise, and cannot be breast-feeding as patients must be receiving cytotoxic chemotherapy, during which breast-feeding is contraindicated
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Patients cannot have documentation in the medical record of current alcohol or substance abuse
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Engaged in full time gainful employment of at least 30 hours per week at the time of cancer diagnosis
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Currently no self-report of engagement in competitive sports (e.g. not training for running races, triathlons, etc) AND no self-report of twice weekly progressive resistance exercise training within the past year
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Self-reported ability to walk for 6 minutes (use of assistive devices will be allowed)
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Not participating in another weight loss, physical activity, or dietary intervention clinical trial
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Predicted 6MWT distance of 450 meters or less
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Concurrent enrollment in treatment or supportive care trials (other than those focused on weight loss or exercise) is allowed with the permission of the Alliance Executive Officer and both studies' study chairs
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Eligibility is restricted to individuals who can comprehend and read English given that participation in the study will require the ability to read intervention materials and work with a coach through telehealth sessions
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): The trial is unable to accommodate the needs of deaf or blind participants as the study relies on language and visualization of exercise through telehealth sessions
* CLINICAL STAKEHOLDER ELIGIBILITY CRITERIA: Clinicians and research staff from enrolling sites who meet following criterion will be deemed eligible to participate as a clinical stakeholder:

  * Providing clinical care for participating patients on this study
* CLINICAL STAKEHOLDER ELIGIBILITY CRITERIA: Ability to speak and understand English

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-02-18 (Estimated)

PRIMARY OUTCOMES:
Percentage of completed exercise sessions (Feasibility) | Up to 6 months
  Feasibility will be defined through intervention adherence. Will set a priori thresholds for this outcome to define success as detailed. For evaluating the uptake of the intervention, will assess the percentage of enrolled participants who complete at least 70% of prescribed exercise sessions. Will calculate the proportion of participants meeting this threshold and compare it to the predefined success criterion of 80%. Descriptive statistics (percentages) will be reported along with 95% confidence intervals.
Intervention attrition rate (Feasibility) | Up to 6 months
  Feasibility will be defined through intervention attrition. Will set a priori thresholds for this outcome to define success as detailed. To examine attrition from the trial, will calculate the attrition rate by dividing the number of participants who drop out of the trial by the total number of enrolled participants. The a priori acceptable attrition rate is no greater than 20%. Descriptive statistics (attrition rate) will be presented, and a comparison with the predefined threshold will be made.

SECONDARY OUTCOMES:
Weekly recruitment rate | From the date that the study is activated at all 4 enrolling sites and the first patient is enrolled, assessed up to 58 weeks
  Feasibility of enrolling a diverse patient population will be defined by: Enrolling 80 patients over a 58-week time period, from the date that the study is activated at all 4 enrolling sites and the first patient is enrolled. Descriptive statistics (mean, standard deviation) will be reported for weekly recruitment, along with graphical representations of recruitment trends over time.
Retaining a diverse patient population | From the date that the study is activated at all 4 enrolling sites and the first patient is enrolled, assessed up to 58 weeks
  Descriptive statistics (percentages) will be summarized for patients who meet at least one of the following criteria: Racial or ethnic minority status (African American, Hispanic, Native American, Pacific Islander), low socioeconomic status (defined as residing in an area in one of the top two quintiles of the Neighborhood Deprivation Index), residing in a rural area (Rural-Urban Continuum Codes or Rural-Urban Commuting Area Code, code 4-10).

OTHER OUTCOMES:
Change in 6 Minute Walk Test (6MWT) distance | From baseline to end of intervention, which is defined as end of chemotherapy (within 4 weeks of the final chemotherapy administration) or up to a total of 6 months of intervention, whichever comes first
  Descriptive statistics (mean, standard deviation) will be used to summarize changes in 6MWT distance in the study population between baseline and the post-intervention time point.
Change in grip strength | From baseline to end of intervention, which is defined as end of chemotherapy (within 4 weeks of the final chemotherapy administration) or up to a total of 6 months of intervention, whichever comes first
  Descriptive statistics (mean, standard deviation) will be used to summarize changes in grip strength in the study population between baseline and the post-intervention time point
Objective changes in physical activity | From baseline to end of intervention, which is defined as end of chemotherapy (within 4 weeks of the final chemotherapy administration) or up to a total of 6 months of intervention, whichever comes first
  Descriptive statistics (mean, standard deviation) will be used to summarize changes in objectively measured physical activity using the accelerometer, including average daily step count, average daily minutes of sedentary time, light activity, and moderate-to-vigorous activity.
Self-reported changes in physical activity | From baseline to end of intervention, which is defined as end of chemotherapy (within 4 weeks of the final chemotherapy administration) or up to a total of 6 months of intervention, whichever comes first
  Descriptive statistics (mean, standard deviation) will be used to summarize self-reported changes (7-Day Physical Activity Recall Interview) in physical activity in the study population between baseline and the post-intervention time point.
Relationship between predicted 6MWT and baseline 6MWT | At baseline
  Person correlation coefficient will be used to summarize the relationship between the predicted 6MWT and the baseline 6MWT.
Changes in patient reported outcomes | From baseline to end of intervention, which is defined as end of chemotherapy (within 4 weeks of the final chemotherapy administration) or up to a total of 6 months of intervention, whichever comes first
  Descriptive statistics (mean, standard deviation) will be used to summarize changes in patient reported outcomes between baseline, end of intervention, and 3-months post intervention in the study population.
Employment status | Up to 3-months post-intervention
  Descriptive statistics (frequency table) histogram will be used to explore the employment status over time in the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ligibel, MD, Study Chair — Alliance for Clinical Trials in Oncology; Kathryn Schmitz, MD, Study Chair — Alliance for Clinical Trials in Oncology

IPD SHARING:
Plan to Share IPD: Undecided